CLINICAL TRIAL: NCT03611452
Title: Simple Continuous, Subcuticular and Interrupted Skin Suturing of Episiotomy and 2nd-degree Perineal Tears : A Comparative Study
Brief Title: Simple Continuous, Subcuticular and Interrupted Skin Suturing of Episiotomy and 2nd-degree Perineal Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCIE
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Episiotomy Wound
MeSH Terms: interventions — Episiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simple continuous (Experimental): the sutures will be taken continuously by simple method
  Interventions: Procedure: Episiotomy
- subcuticular (Active Comparator): the sutures will be taken subcuticular
  Interventions: Procedure: Episiotomy
- interrupted (Active Comparator): the sutures will be taken interrupted method
  Interventions: Procedure: Episiotomy

INTERVENTIONS:
Procedure: Episiotomy — repair of perineal muscles and skin

SUMMARY:
Millions of women worldwide undergo perineal suturing after childbirth and the type of repair may have an impact on pain and healing.

The skin as a barrier between the internal structures and the external environment is exceptionally susceptible to injury, either through accidental injury or planned surgical incision. Today, as surgery increases in complexity, and the heightened public awareness of scar cosmesis and skin healing need to be optimized to ensure the overall success of the surgical procedure

ELIGIBILITY:
Inclusion Criteria:

* Normal vaginal delivery.
* At term (37 40 weeks ).
* Live baby.
* Vertex presentation

Exclusion Criteria:

* Third and fourth degree perineal tear.
* Instrumental vaginal delivery.
* Previous perineal surgery.
* Anaemia with hemoglobin level < 9 g/dl.
* Diabetes mellitus.
* Coagulation abnormalities.
* Postpartum hemorrhage.
* Delivery conducted outside Woman HealthHospital.
* Breech delivery.
* Body mass index >35 kg/m2.
* Local infectious lesions.
* Anal fissures or hemorrhoid.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
the mean score of Perineal pain during vaginal suturing | 10 minutes
  assessment through visual analog scale score from 0 - 10 at every step of repair